CLINICAL TRIAL: NCT05782270
Title: Comparison of Antithrombotic Therapy After Coronary Artery Bypass Grafting Combined With Coronary Endarterectomy
Brief Title: Antithrombotic Therapy After Coronary Artery Bypass Grafting Combined With Coronary Endarterectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-GSP-QN-11
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anticoagulation; Coronary Endarterectomy
Keywords: coronary endarterectomy; coronary artery bypass grafting; anticoagulation; antiplatelet
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAPT (Other): Comparison group: dual antiplatelet only
  Interventions: Drug: DAPT; Other: CE+CABG
- DAPT+warfarin (Experimental): Intervention group: dual antiplatelet combined with warfarin
  Interventions: Drug: Warfarin; Drug: DAPT; Other: CE+CABG

INTERVENTIONS:
Drug: Warfarin — dual antiplatelet therapy combined with warfarin
  Arms: DAPT+warfarin
Drug: DAPT — Dual antiplatelet therapy (aspirin plus either clopidogrel or ticagrelor)
Other: CE+CABG — Coronary endarterectomy combined with coronary artery bypass grafting

SUMMARY:
Coronary endarterectomy (CE) combined with coronary artery bypass grafting (CABG) can be the final option for achieving complete revascularization in diffuse coronary artery disease patients. Since the exposure of subendothelial tissue to the blood flow after CE, the coagulation cascade can be activated, resulting in the increased risk of graft failure. Therefore, anticoagulation with warfarin in this group of patients might be beneficial. However, evidence is limited. This study aims to compare the clinical outcomes between dual antiplatelet therapy with or without warfarin after CE+CABG.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diffuse coronary artery disease undergoing CE+CABG during the study period.
* No contraindications for both dual antiplatelet therapy and anticoagulation therapy with warfarin.
* Must be able to swallow tablets after the surgery.

Exclusion Criteria:

1. Patients with high bleeding risk (HAS-BLED ≥ 3);
2. Patients undergoing concomitant aortic valve or mitral valve surgery, or undergoing cardiac surgery for the second time;
3. Emergency surgery;
4. Serum creatinine >130μmol/L, or significant liver dysfunction (elevated ALT and/or AST);
5. History of digestive or urinary tract bleeding, active gastric bleeding caused by gastric ulcer, or postoperative new-onset gastric bleeding;
6. History of hemorrhagic stroke, or platelet dysfunction;
7. Allergic or with contraindication to any of aspirin, clopidogrel or warfarin;
8. Participated in other clinical trial for drug or device within 30 days;
9. Pregnant or planning to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of coronary endarterectomy-targeted graft patency. | 6 months postoperatively
  Defined as less than 50% stenosis of the coronary endarterectomy target and coronary endarterectomy-targeted graft evaluated through either of coronary computed tomography angiography or coronary angiography.

SECONDARY OUTCOMES:
Number of patients suffering from major adverse cardiovascular and cerebrovascular events | During 6-month follow-up
  Major adverse cardiovascular and cerebrovascular events is defined as the composite of all-cause death, myocardial infarction, stroke and repeat revascularization.
Bleeding events | during 6-month follow-up
  The Bleeding Academic Research Consortium (BARC) scale type 2~5 [see in reference].

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Derived] Tiemuerniyazi X, Yang Z, Yang E, He L, Chen L, Huang S, Nan Y, Song Y, Xu F, Yuan X, Hu Z, Zhao W, Feng W. Postoperative antithrombotic therapy after coronary artery bypass grafting combined with coronary endarterectomy (PATH-CARE): study protocol for a randomised controlled clinical trial. BMJ Open. 2025 Nov 9;15(11):e104950. doi: 10.1136/bmjopen-2025-104950. PMID 41213699